CLINICAL TRIAL: NCT03636243
Title: Comparative Evaluation of the Evolution of Arterial and Microcirculatory Endothelial Function in Obese Patients With Type-2 Diabetes Versus Non-diabetic Obese Patients After a First Bariatric Surgery
Acronym: BariVaDia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-02/APM-01
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery; Obese; Type2 Diabetes
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of obese patients with type-2 diabetes (Other)
  Interventions: Biological: Vascularly biological assessment; Biological: Analysis of vasomotor endothelial function; Biological: Analysis of arterial compliance; Biological: Exploration of microcirculation; Biological: Venous Doppler Ultrasound; Biological: Arterial pressure measurement; Biological: Intima-Media Thickness measurement; Biological: Exploration of neuropathy; Behavioral: level of physical activity
- Group of non-diabetic obese patients (Other)
  Interventions: Biological: Vascularly biological assessment; Biological: Analysis of vasomotor endothelial function; Biological: Analysis of arterial compliance; Biological: Exploration of microcirculation; Biological: Venous Doppler Ultrasound; Biological: Arterial pressure measurement; Biological: Intima-Media Thickness measurement; Biological: Exploration of neuropathy; Behavioral: level of physical activity; Other: thoracic scanner

INTERVENTIONS:
Biological: Vascularly biological assessment — 22.5 ml of blood will be collected at day -15, month 3 and month 12.
Biological: Analysis of vasomotor endothelial function — Evaluation of the peripheral endothelial function by digital tonometry using the 'EndoPATTM2000' system [Itamar Medical Ltd., Caeserea, Israel] before and after induction of post occlusive reactive hyperemia at day -15, month 3 and month 12.
Biological: Analysis of arterial compliance — Evaluation of the aortic pulse wave velocity in the aortofemoral segment or in the periphery (on the arm-ankle segment) by calculation of central aortic pressure (CAP) using the tonometric system 'Complior ™' [Alam Medical, France] at day -15, month 3 and month 12
Biological: Exploration of microcirculation — The microcirculation exploration via analysis of the curves recorded by Laser Doppler at day -15, month 3 and month 12
Biological: Venous Doppler Ultrasound — aneurysm screening at day -15, month 3 and month 12
Biological: Arterial pressure measurement — measurement of the systolic pressure at the toe using the SysToe™ device, and measurement of systolic and diastolic blood pressure using the Dinamap™ device at day -15, month 3 and month 12
Biological: Intima-Media Thickness measurement — Intima-Media Thickness measurement using an ultrasound machine at day -15, month 3 and month 12
Biological: Exploration of neuropathy — non-invasive measurement of sudomotor function by SUDOSCAN at day -15, month 3 and month 12
Behavioral: level of physical activity — pedometer collecting the number of steps during the four days before visits at day -15, month 3 and month 12
Other: thoracic scanner — non-injected thoracic scanner visit at month 3
  Arms: Group of non-diabetic obese patients

SUMMARY:
The weight reduction obtained after a first bariatric surgery would improve the vascular (correction of endothelial dysfunction, improvement of arterial wall compliance and evolution of the atherothrombotic process) and microcirculatory function in obese patients with type-2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years old and under 70 years old
* The patient is available for a follow-up of 12 months
* The patient signed the consent form
* The patient must be affiliated or beneficiary to an health care plan
* The patient is followed in hospital day care in the endocrine and metabolic disorders department at Nimes University Hospital for a first bariatric surgery

Exclusion Criteria:

* The subject participates in another interventional study.
* The subject is in an exclusion period determined by a previous study.
* The subject is under the protection of justice, guardianship or curatorship.
* The subject refuses to sign the consent.
* It is not possible to give the subject informed information.
* The patient is pregnant or breastfeeding.
* Subject with known advanced atherothrombotic disease (arterial disease of the lower limbs, significant carotid plaque (generating stenosis> 50%), history of myocardial infarction, stroke)
* The subject is type 1 diabetic.
* The subject has already had a bariatric surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) | day -15
  Measured to the finger by tonometry using the "Endo-Pat 2000 device"
Reactive Hyperemia Index (RHI) | Month 3
  Measured to the finger by tonometry using the "Endo-Pat 2000 device"

SECONDARY OUTCOMES:
Reactive Hyperemia Index (RHI) | day -15, Month 12
  reactive hyperemia index (%)
Compare the concentration of the vascular endothelial growth factor marker of endothelial function in both groups and between groups | day -15
  pg/mL
Compare the concentration of the vascular endothelial growth factor marker of endothelial function in both groups and between groups | Month 3
  pg/mL
Compare the concentration of the vascular endothelial growth factor marker of endothelial function in both groups and between groups | Month 12
  pg/mL
Compare the concentration of the soluble fms-like tyrosine kinase-1 markers of endothelial function in both groups and between groups | Day -15
  pg/mL
Compare the concentration of the soluble fms-like tyrosine kinase-1 markers of endothelial function in both groups and between groups | Month 3
  pg/mL
Compare the concentration of the soluble fms-like tyrosine kinase-1 markers of endothelial function in both groups and between groups | Month 12
  pg/mL
Compare the concentration of the fibrinogen marker of endothelial function in both groups and between groups | Day -15
  g/L
Compare the concentration of the fibrinogen marker of endothelial function in both groups and between groups | Month 3
  g/L
Compare the concentration of the fibrinogen marker of endothelial function in both groups and between groups | Month 12
  g/L
Compare the concentration of the D-dimer marker of endothelial function in both groups and between groups | Day -15
  ng/ml
Compare the concentration of the D-dimer marker of endothelial function in both groups and between groups | Month 3
  ng/ml
Compare the concentration of the D-dimer marker of endothelial function in both groups and between groups | Month 12
  ng/ml
Evaluate the physical activity | Day -15
  number of steps in previous 4 days
Evaluate the physical activity | Month 3
  number of steps in previous 4 days
Evaluate the physical activity | Month 12
  number of steps in previous 4 days
Creation of a biobank | Day -15
  storage of blood sample
Creation of a biobank | Month 3
  storage of blood sample
Creation of a biobank | Month 12
  storage of blood sample
Compare toe pressure using the SysToe device in both groups and between groups | Day -15
  mmHg
Compare toe pressure using the SysToe device in both groups and between groups | Month 3
  mmHg
Compare toe pressure using the SysToe device in both groups and between groups | Month 12
  mmHg
Compare the sweat function using the" Sudoscan" device in both groups and between groups | Day -15
  µV
Compare the sweat function using the "Sudoscan" device in both groups and between groups | Month 3
  µV
Compare the sweat function using the "Sudoscan" device in both groups and between groups | Month 12
  µV
Compare the vibratory sensitivity using a neurothesiometer in both groups and between groups | Day -15
  Hz
Compare the vibratory sensitivity using a neurothesiometer in both groups and between groups | Month 3
  Hz
Compare the vibratory sensitivity using a neurothesiometer in both groups and between groups | Month 12
  Hz
Compare the sensitive conduction velocity in both groups and between groups | Day -15
  m/s
Compare the sensitive conduction velocity in both groups and between groups | Month 3
  m/s
Compare the sensitive conduction velocity in both groups and between groups | Month 12
  m/s
Evaluate the presence of neuropathic pain using the questionnaire "Neuropathic Pain in 4 Questions" | Day -15
  If the score is greater than or equal to 4, the test is positive.
Evaluate the presence of neuropathic pain using the questionnaire "Neuropathic Pain in 4 Questions" | Month 3
  If the score is greater than or equal to 4, the test is positive.
Evaluate the presence of neuropathic pain using the questionnaire "Neuropathic Pain in 4 Questions" | Month 12
  If the score is greater than or equal to 4, the test is positive.
Evaluate the quality of life using the "Quality Of Life, Obesity and Dietetics" questionnaire | Day -15
  It has 36 items, rated from 1 (always / enormously) to 5 (never / not at all). It explores five dimensions (physical impact - Q1-Q11, psychosocial impact - Q12-Q22, impact on sex life - Q23-Q26, nutritional well-being - Q27-Q31 and diet experience - Q32-Q36). The rating of each dimension is reported at 100. The higher the score is close to 100, the better the quality of life related to this dimension.
Evaluate the quality of life using the "Quality Of Life, Obesity and Dietetics" questionnaire | Month 3
  It has 36 items, rated from 1 (always / enormously) to 5 (never / not at all). It explores five dimensions (physical impact - Q1-Q11, psychosocial impact - Q12-Q22, impact on sex life - Q23-Q26, nutritional well-being - Q27-Q31 and diet experience - Q32-Q36). The rating of each dimension is reported at 100. The higher the score is close to 100, the better the quality of life related to this dimension.
Evaluate the quality of life using the "Quality Of Life, Obesity and Dietetics" questionnaire | Month 12
  It has 36 items, rated from 1 (always / enormously) to 5 (never / not at all). It explores five dimensions (physical impact - Q1-Q11, psychosocial impact - Q12-Q22, impact on sex life - Q23-Q26, nutritional well-being - Q27-Q31 and diet experience - Q32-Q36). The rating of each dimension is reported at 100. The higher the score is close to 100, the better the quality of life related to this dimension.
Analysis of post-ischemic hyperemia using the laser doppler Perimed. | Day -15
Analysis of post-ischemic hyperemia using the laser doppler Perimed. | Month 3
Analysis of post-ischemic hyperemia using the laser doppler Perimed. | Month 12
Analysis of cutaneous vasomotion using the laser doppler Perimed. | Day -15
Analysis of cutaneous vasomotion using the laser doppler Perimed. | Month 3
Analysis of cutaneous vasomotion using the laser doppler Perimed. | Month 12
study of the peri-aortic and peri-brachial adipose tissue (TAPV) | Month 3
  comparison of peri-aortic and peri-brachial peri-vascular adipose tissue (PVAPT), before and 3 months after CB, in the group of 20 non-diabetic obese patients. Semi-automatic quantification with identification by the density of the pixels corresponding to the TA (-195 to -45 HU (Hounsfield Units) and 3D reconstruction for volumetric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Antonia PEREZ-MARTIN, Pr, Principal Investigator — Nîmes University Hospital
Locations (1):
- CHU Nimes, Nîmes, France